CLINICAL TRIAL: NCT00325793
Title: An Open-Label Prospective Study to Evaluate the Safety and Efficacy of Double or Triple Concentrated Intravenous Nicardipine for Treatment of Hypertension in Patients With Ischemic Stroke, Intracerebral Hemorrhage or Subarachnoid Hemorrhage
Brief Title: IV Double and Triple Concentrated Nicardipine for Stroke and ICH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OSF Healthcare System (Other)
Collaborators: PDL BioPharma, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0012003
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2006-05

CONDITIONS: Hypertension
Keywords: nicardipine; hypertension; intracerebral hemorrhage; ischemic stroke
MeSH Terms: conditions — Hypertension; Cerebral Hemorrhage; Ischemic Stroke | interventions — Nicardipine

INTERVENTIONS:
Drug: Nicardipine

SUMMARY:
Hypertension (high blood pressure) can often cause neurological worsening in patients with stroke, intracerebral hemorrhage and subarachnoid hemorrhage. Intravenous infusion of nicardipine (Cardene) for control of hypertension is FDA approved. The disadvantage of Nicardipine IV drip is the relative large volume of fluid needed (up to 150 cc/hr). The purpose of this study is to evaluate safety and efficacy of double or triple concentrated peripheral intravenous (IV) Nicardipine.

DETAILED DESCRIPTION:
Hypertension can often cause neurological worsening in patients with either ICH or SAH. Hypertension has been related to increased incidence of intracranial hemorrhage in patients who are treated with thrombolytics or on anticoagulation. Timely control of hypertension is directly related to the outcome of these patients. Furthermore, unlike in the conditions of hypertensive emergency or urgency, gentle titration to control the blood pressure is recommended in patients with either ischemic cerebral infarction or hemorrhage. Therefore the ideal agent to control hypertension in these patients would have these characteristics:

* Rapid onset of action
* Predictable dose response
* Titratable to desired BP
* Minimal dosage adjustments
* Minimal adverse effects
* No increase in INTRACRANIAL PRESSURE (ICP)
* Easy transition to oral formulation for long-term maintenance

Currently, only IV sodium nitroprusside, nitroglycerine, enalapril and esmolol are used for controlling blood pressure in patients with IS, ICH and SAH. These agents are difficult to titrate and may potentially be harmful to brain cells.

Nicardipine offers several advantages in blood pressure control. It may cause dilatation of the coronary vessels while has no effect on cardiac conduction. It is not associated with coronary steal. As the only IV calcium channel blocker approved for the treatment of hypertension, nicardipine is vasoselective, and has a rapid onset and precisely controllable in a variety of patient types. It is as effective as sodium nitroprusside with fewer dose adjustments. It has documented safety with a low incidence of side effects. It requires minimal dose adjustments.

The disadvantage of Nicardipine IV drip is the relative large volume of fluid needed (up to 150 cc/hr). In patients with ischemic cerebral stroke (IS) or hemorrhage (ICH), intravenous infusion of large volume can contribute to cerebral edema or increase in intracranial pressure (ICP). If the infusion of nicardipine can be double or triple concentrated without the need of a central line, it not only offers titratable BP control, but also less overall volume to infuse the drug.

This is a phase IV prospective, open-label, dose regimen study of double or triple concentration nicardipine infusion for controlling blood pressure in patients with either ischemic cerebral infarction (IS) or intracerebral hemorrhage (ICH) or subarachnoid hemorrhage (SAH). Once the patient has the need for rapid control of blood pressure, he or she will be eligible for the study. The first 25 patients will be consented for the double dose treatment and the next 25 patients will be consented for the triple dose treatment. The patient will be followed during the infusion period for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 years of age or older.
* Acute ischemic cerebral stroke (IS) with uncontrollable hypertension that may need to be controlled for the purpose of considering thrombolytic therapy or anticoagulation therapy.
* Intracerebral hemorrhagic (ICH) stroke patients, including subarachnoid hemorrhage (SAH) (surgically treated or not), any territory with an appropriate study (head CT scan or MRI scan) providing results consistent with this diagnosis, who may require the control of hypertension or control of blood pressure.

Exclusion Criteria:

* Allergy to Nicardipine or known hypersensitivity to Nicardipine.
* Chronic renal failure or Creatinine blood sample levels> 2.0.
* Impaired hepatic function defined as a two times value of liver enzymes.
* Severe left ventricular dysfunction defined as ventricular ejection fraction < 30%.
* Patients or authorized representative who refused be enrolled into this study.
* Advanced aortic stenosis.
* Pregnant or nursing women will not be enrolled in this study.
* No patient will be allowed to be enrolled in this study more than once.
* Patients may not be enrolled into other clinical studies during their involvement with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-01

PRIMARY OUTCOMES:
• Demonstrate the feasibility and safety of double and triple concentrated peripheral intravenous Nicardipine for patients in the Neuroscience Critical Care Unit.

SECONDARY OUTCOMES:
Time and dosage adjustment needed to reach the target BP range
Safety
To evaluate the tolerance of the double or triple concentrated Nicardipine

CONTACTS AND LOCATIONS:
Overall Officials: David Wang, DO, Principal Investigator — OSF Stroke Center
Locations (1):
- OSF Stroke Center, Peoria, Illinois, United States